CLINICAL TRIAL: NCT07382479
Title: A Prospective, International, Multi-center, Interventional Trial of Advanced Epithelial Ovarian Cancer Patients Offered Three Cycles of Neoadjuvant Chemotherapy (NACT) and Triaged With KELIM Score. Patients With Favorable Score Will Undergo Interval Debulking Surgery (IDS) Followed by Another 3 Cycles of NACT, While Those With Unfavorable Will Undergo Another 3 Cycles of NACT Followed by Delayed Interval Debulking Surgery (DIDS).
Brief Title: NeoAdjuvant ChemoTherapy With KELIM Guided Interval vs. Delayed Interval Debulking Surgery
Acronym: NACT-KELIM ID
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aristotle University Of Thessaloniki (Other)
Responsible Party: Principal Investigator, Dimitrios Zouzoulas, Gynecological Oncologist, MSc, PhD, FEBS-BS, Aristotle University Of Thessaloniki
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022-Β2015-230
Record Dates: First submitted 2026-01-27; First posted 2026-02-02 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Intervention Model Description: * ARM A: 3 cycles of NACT with a favorable KELIM score will undergo IDS followed by 3 cycles of NACT
  * ARM B: 3 cycles of NACT with an unfavorable KELIM score will undergo 3 more cycles of NACT followed by DIDS
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ARM A: IDS (Active Comparator): 3 cycles of NACT with a favorable KELIM score underwent IDS followed by 3 cycles of NACT
  Interventions: Procedure: 3 cycles of NACT with favorable KELIM score will undergo IDS followed by 3 cycles of NACT
- ARM B: DIDS (Experimental): 3 cycles of NACT with an unfavorable KELIM score will undergo 3 cycles of NACT followed by DIDS
  Interventions: Procedure: 3 cycles of NACT with unfavorable KELIM score will receive 3 more cycles of NACT followed by DIDS

INTERVENTIONS:
Procedure: 3 cycles of NACT with unfavorable KELIM score will receive 3 more cycles of NACT followed by DIDS — 3 cycles of NACT with unfavorable KELIM score will receive 3 more cycles of NACT followed by DIDS
  Arms: ARM B: DIDS
Procedure: 3 cycles of NACT with favorable KELIM score will undergo IDS followed by 3 cycles of NACT — 3 cycles of NACT with favorable KELIM score will undergo IDS followed by 3 cycles of NACT
  Arms: ARM A: IDS

SUMMARY:
A prospective, international, multi-center, interventional trial of advanced epithelial ovarian cancer patients offered three cycles of neoadjuvant chemotherapy (NACT) and triaged with KELIM score. Patients with favorable score will undergo interval debulking surgery (IDS) followed by another 3 cycles, while those with unfavorable score will undergo another 3 cycles of NACT followed by delayed interval debulking surgery (DIDS).

DETAILED DESCRIPTION:
Primary debulking surgery (PDS) followed by adjuvant chemotherapy is the cornerstone of advanced ovarian cancer treatment. However, frail patients, patients with high tumor burden in the upper abdomen or extra-abdominal metastases may benefit from neoadjuvant chemotherapy (NACT) followed by interval debulking surgery (IDS). In recent years, three randomized non-inferiority trials have demonstrated that NACT is a valid alternative to PDS. Similarly, the preliminary results from the TRUST trial showed that the primary endpoint of overall survival (OS) was not met, with numerical longer OS in PDS group compared to NACT in non-frail ovarian cancer patients. The optimal number of NACT cycles has not yet been established. Most studies in the literature recommend 3-4 cycles. However, in real-world clinical practice some patients receive more than 5 cycles before surgery, so delayed interval debulking surgery (DIDS) is proposed as an alternative. The rationale is to allow for maximal tumor shrinkage and improved likelihood of complete gross resection, while reducing perioperative morbidity. Retrospective data show that DIDS may be considered as an alternative for advanced ovarian cancer patients with a high tumor burden, when complete gross resection cannot be achieved during IDS.

Furthermore, the success of the above-mentioned treatment plans depends on tumor chemosensitivity and the ability to achieve complete gross resection, because residual disease after cytoreduction remains the most important prognostic factor. On the other hand, 15-20% of patients with advanced ovarian cancer will be poor responders to chemotherapy, so there is the need for accurate non-invasive chemo-sensitivity predictors to guide treatment decisions in the first-line setting, which is acknowledged by ESGO and ESMO. Monitoring of CA-125 decline during chemotherapy for the prediction of treatment response (13) and as a way to overcome imaging limitations, has been one of the main points of research in ovarian cancer patients. The ELIMination rate constant K (KELIM), a modeled kinetic parameter based on CA-125 measurements during the first 100 days of systemic therapy (adjuvant of neoadjuvant chemotherapy), has emerged as a valuable predictor. It is a mathematical modeling method based not on absolute values of the biomarker, but on the longitudinal kinetics (CA-125 elimination) during treatment, completely independent of renal function. Retrospective data show that KELIM score is an independent prognostic biomarker for survival outcomes, that can predict chemosensitivity, and that can safely triage patients undergoing NACT and guide who will benefit from IDS and DIDS, respectively.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 - 85 years old
* Histologically proven epithelial ovarian cancer, fallopian tube carcinoma, or primary peritoneal carcinoma, high grade serous or endometrioid
* ECOG Performance status 0 - 1
* Documented International Federation of Gynecologic Oncology (FIGO) 2014 stage IIIB, IIIC or IVA unfit and/or with unresectable disease for complete primary debulking surgery (preferably triaged by "Fagotti" diagnostic laparoscopy)
* HIPEC is an option after IDS or DIDS
* Sufficiently good bone marrow, liver, and renal function to receive chemotherapy and subsequently undergo surgery

Exclusion Criteria:

* Pregnancy
* Synchronous malignancies at the time of diagnosis or in the 3 years prior to starting the study treatment
* Comorbidities that may contraindicate surgery or chemotherapy as planned per protocol
* Mucinous, clear-cell, carcinosarcoma or low-grade serous adenocarcinoma histological subtypes
* Stable disease or progression of disease (preferably triaged by "Fagotti" diagnostic laparoscopy) after 6 cycles of NACT, before DIDS.

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 485 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2031-04-01 (Estimated); Study Completion 2034-04-01 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | After 5 years from last patient enrollment

SECONDARY OUTCOMES:
Progression free survival (PFS) | After 2 years from last patient enrollment.
Complete gross resection rate (residual disease: 0 cm) | After a month from cytoreduction
Postoperative complications (Clavien-Dindo classification) | After a month after cytoreduction
  Postoperative complications will be graded using the Clavien-Dindo classification of surgical complications, which ranges from Grade I to Grade V, with higher grades indicating more severe complications and Grade V representing death
Quality of life (QoL) (EORTC QLQ-C30 questionnaire) | After a month from cytoreduction
  Health-related quality of life will be assessed with the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30), scored from 0 to 100. For the global health and functional scales, higher scores indicate better functioning/quality of life, whereas for symptom scales higher scores indicate greater symptom burden (worse outcome)

CONTACTS AND LOCATIONS:
Overall Officials: Dimitrios Tsolakidis, Dr.Prof., Principal Investigator — Artistotle University of Thessaloniki

IPD SHARING:
Plan to Share IPD: No
Sharing of IPD only after contact with the principal investigator for the synthesis of future studies.

REFERENCES:
- [Background] Zouzoulas D, Tsolakidis D, Tzitzis P, Sofianou I, Chatzistamatiou K, Theodoulidis V, Topalidou M, Timotheadou E, Grimbizis G. The Use of CA-125 KELIM to Identify Which Patients Can Achieve Complete Cytoreduction after Neoadjuvant Chemotherapy in High-Grade Serous Advanced Ovarian Cancer. Cancers (Basel). 2024 Mar 24;16(7):1266. doi: 10.3390/cancers16071266. PMID 38610943
- [Background] Zouzoulas D, Sofianou I, Tzitzis P, Theodoulidis V, Chatzistamatiou K, Timotheadou E, Grimbizis G, Tsolakidis D. The Role of Delayed Interval Debulking Surgery (DIDS) in the Surgical Treatment of Advanced Epithelial Ovarian Cancer: A Retrospective Cohort from an ESGO-Certified Center. Med Sci (Basel). 2025 Oct 2;13(4):217. doi: 10.3390/medsci13040217. PMID 41133497